CLINICAL TRIAL: NCT03167216
Title: Mast Cells in Male Pelvic Pain and and Lower Urinary Tract Dysfunction
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Praveen Thumbikat, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00202831; R01DK083609 (NIH)
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome
Keywords: chronic pain; prostatitis; pelvic pain
MeSH Terms: conditions — Prostatitis; Chronic Pain; Pelvic Pain | interventions — Cromolyn Sodium; Cetirizine

STUDY DESIGN:
Intervention Model Description: Comparison of mast cell tryptase levels and changes in symptom scores after treatment with cromolyn sodium and cetirizine hydrochloride
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment arm (Experimental): Treated arm with cromolyn sodium and cetirizine hydrochloride
  Interventions: Drug: Cromolyn Sodium; Drug: Cetirizine Hydrochloride

INTERVENTIONS:
Drug: Cromolyn Sodium — Mast cell stabilizer
  Other Names: Gastrocrom
Drug: Cetirizine Hydrochloride — Histamine receptor antagonist
  Other Names: Zyrtec

SUMMARY:
The objective of this study is to evaluate inhibition of mast cells and the histamine 1 receptor (H1R) for treatment of chronic prostatitis (CP) and chronic pelvic pain syndrome (CPPS).

DETAILED DESCRIPTION:
Chronic pelvic pain is a hallmark of patients with CPPS, a non-bacterial category of prostatitis that is a significant source of morbidity in men. The cause of CPPS is unknown and there is a lack of biomarkers for diagnosis of this syndrome. Research in animal models of CP/CPPS have pointed to a role for mast cells and their degranulation constituents including mast cell tryptase in the development of pelvic pain and lower urinary tract symptoms. This study aims to evaluate the ability of FDA approved and marketed drugs to inhibit the release of mast cell tryptase and to ameliorate symptoms in patients with CP/CPPS.

This is an open label study to evaluate the efficacy of Cromolyn Sodium Oral Solution and Cetirizine hydrochloride (tablet) in men with CP/CPPS to reduce mast cell tryptase levels in expressed prostatic fluids and to show improvement in symptoms of CP/CPPS. There is no control group for the study. The difference between pre- and post-treatment levels across individuals will be assessed.

The study will consist of 3 periods: the Screening Period (Days -7 to -1), the Treatment Period (Days 1 to 21), and the Follow-up Period (7 days) after the last dose at Day 21.

During screening, subjects will be admitted to the clinic, undergo specimen (Expressed prostatic secretions (EPS), urine and blood) collection and recording of their baseline questionnaire responses Subjects will provide a basic health history, including current general health, adverse events, medications or treatments within the past 5 years. A physical examination including vital heart rate, breathing rate, blood pressure, temperature, height, weight and body mass will be taken. Subsequently, EPS from eligible subjects will be collected by the clinical team and assayed for the levels of mast cell tryptase within 24 hours of sample collection at the screening visit. 20 subjects with elevated mast cell tryptase will be identified and will be eligible for receiving the study medication from the Investigational pharmacy at Northwestern University.

Eligible subjects will be required to take medication for days 1-21 (Week 1-3), record their symptom scores weekly using the NIH-CPSI, and record all safety related symptoms.

Subjects will return to the clinic after the completion of three weeks of treatment. Expressed prostatic secretions (EPS), blood as well as a voided bladder 1, 2 and 3 (VB1-3) urine specimens will be collected as at baseline and after the last dose at day 21 for evaluating mast cell tryptase levels. A review subject's general health, adverse events, and any medications that have changed since the last visit will be collected. Vital signs (heart rate, breathing rate, blood pressure, temperature, weight and BMI will be collected.

Treated subjects will be contacted by phone 7 days after treatment by the study coordinator to follow up on any study related adverse effects or changes in symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male ages 21-80 years old
* Diagnosed with Category III Chronic Pelvic Pain Syndrome
* Patients reporting pain or discomfort in any of the 8 domains of the NIH_ Chronic Prostatitis Symptom Index (NIH-CPSI).
* CP/CPPS symptoms must have been present for the majority of the time during any 3 months in the previous 6 months.
* Mast cell tryptase levels in EPS above a control threshold of 25ng/ml based on healthy men.

Exclusion Criteria:

* Females
* Males <21 and >80 years old
* Patients with a known hypersensitivity to cromolyn sodium or cetirizine hydrochloride
* Patients with impaired renal or hepatic function.
* Mast cell tryptase levels in EPS equal to or below a control threshold of 25ng/ml based on healthy men.

Ages: 21 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Mast cell tryptase levels in expressed prostatic secretions | 3 weeks
  Changes in Mast cell tryptase at the end of treatment compared to levels observed before administration of the study drug.

SECONDARY OUTCOMES:
NIH-CPSI score | 3 weeks
  Change in pelvic pain, urinary symptoms and quality of life after treatment
AUA-SI score | 3 weeks
  Change in symptoms of lower urinary tract dysfunction after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Thumbikat, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medical Faculty Foundation, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Done JD, Rudick CN, Quick ML, Schaeffer AJ, Thumbikat P. Role of mast cells in male chronic pelvic pain. J Urol. 2012 Apr;187(4):1473-82. doi: 10.1016/j.juro.2011.11.116. Epub 2012 Feb 17. PMID 22341813
- [Result] Murphy SF, Schaeffer AJ, Thumbikat P. Immune mediators of chronic pelvic pain syndrome. Nat Rev Urol. 2014 May;11(5):259-69. doi: 10.1038/nrurol.2014.63. Epub 2014 Apr 1. PMID 24686526
- [Result] Roman K, Done JD, Schaeffer AJ, Murphy SF, Thumbikat P. Tryptase-PAR2 axis in experimental autoimmune prostatitis, a model for chronic pelvic pain syndrome. Pain. 2014 Jul;155(7):1328-1338. doi: 10.1016/j.pain.2014.04.009. Epub 2014 Apr 13. PMID 24726923